CLINICAL TRIAL: NCT01717248
Title: A Phase 1 Study of Weekly Doses of GCS-100 in Patients With Chronic Kidney Disease
Brief Title: Safety Study of GCS-100 to Treat Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCS-100-CS-4001
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — GCS-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCS-100 (Experimental): GCS-100 will be administered once weekly by a ten minutes injection.
  Interventions: Drug: GCS-100

INTERVENTIONS:
Drug: GCS-100 — GCS-100 is a modified citrus pectin that binds to and sequesteres circulating galectin-3, a protein that has been shown to promote organ disease (fibrosis).

SUMMARY:
The purpose of this study is to evaluate the safety of GCS-100 as a treatment for chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is capable of understanding the purpose and risks of the study and is able to provide written Informed Consent.

  2. Subject is male or female, aged >=18 and <= 75. Patients older than 75 y/o will be included at the request of the investigator and at the discretion of the Medical Monitor .

  3. Adult patients with chronic kidney disease for longer than 12 months and stable in the opinion of the investigator for the past 3 months 4. Systolic blood pressure <=160 mm Hg and >= 90 mm Hg on 2 readings. Diastolic blood pressure <= 100 mm Hg and >= 40 mm Hg on 2 readings during at least one of the screening visits.

  5. Subject is willing to practice birth control. 6. Subject is willing and able to comply with all protocol requirements. 7. Subject has a measureable level of galectin-3 concentration in plasma at any time prior to entry.

  8. Subject has a glomerular filtration rate between 15-45 mL/min/1.73 m2 determined using the CKD-EPI equation (see section 3.6.1) 9. Subject's has clinical laboratory values of:
  1. Hemoglobin ≥9 g/dL
  2. Total bilirubin ≤ 1.5 X Institutional Upper Limit of Normal (IULN)
  3. AST and/or ALT ≤ 2.5 X the upper limit of normal 10. Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least 1 year) and male subjects with partners of childbearing potential must agree to use medically acceptable methods of contraception throughout the study period.

Exclusion Criteria:

1. Subjects who have had treatment with an experimental (unlicensed) drug within 4 weeks or ≤ 5 half-lives prior to treatment with GCS 100.
2. Subjects with kidney disease due to systemic lupus erythematosus (regardless of whether active or in remission), any form of vasculitis (regardless of whether active or in remission), IgA nephropathy, multiple myeloma, polycystic kidney disease, untreated obstructed nephropathy or any other causes that in the opinion of the investigator may put the subject at an increased risk
3. Subject is expected to start renal replacement therapy of any kind within 6 months after enrollment
4. Subjects with previous solid organ transplant
5. Subject is undergoing treatment with immunosuppression agents except for topical agents or inhaled steroids when conditions are chronic and stable.
6. Subject with know history of cancer within the past 5 years prior to enrollment excluding non-melanoma skin cancer that is not being actively treated
7. Subject has a known history of human immunodeficiency virus infection, active hepatitis C, active hepatitis B, or prior history of infection with hepatitis B (HBcAb positive). Medical Monitor may approve if adequate hepatic function has been documented for patients without evidence of cirrhosis for subjects with HCV or prior history of hepatitis B, including, but not limited to liver biopsy.
8. Subject has a clinically relevant active infection and/or a serious co-morbid medical condition such as recent myocardial infarction (within the last 6 months), unstable angina, difficult-to-control congestive heart failure, uncontrolled hypertension, difficult-to-control cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, and/or cirrhosis.
9. Subject had major surgery within 4 weeks prior to Study Day 1.
10. If female, subject is pregnant or breastfeeding.
11. Subject has a concomitant disease or condition, including laboratory abnormalities, which in the opinion of the Investigator could interfere with the conduct of the study or could put the subject at unacceptable risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety | Ongoing
  Assess overall safety of rising dose of GCS-100 in CKD patients

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Pergola, MD, Principal Investigator — Renal Associaties PA, Research Division; Geoffrey Block, MD, Principal Investigator — Denver Nephrologists, PC; Bhupinder Singh, MD, Principal Investigator — Southwest Clinical Research Institute, LLC; George Fadda, MD, Principal Investigator — California Institute of Renal Research
Locations (4):
- United States (4):
  - Southwest Clinical Research Institute, Tempe, Arizona
  - California Institue of Renal Research, La Mesa, California
  - Denver Nephrologists, PC, Denver, Colorado
  - Renal Associates PA / Research Division, San Antonio, Texas